CLINICAL TRIAL: NCT02407431
Title: PaTH Clinical Data Research Network (CDRN) Idiopathic Pulmonary Fibrosis (IPF) Clinician Patient Partnership Cohort
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Temple University (Other); Johns Hopkins University (Other); Penn State University (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Kathleen McTigue, Professor, University of Pittsburgh
Other Study IDs: STUDY20110299; CDRN-1306-04912 (Other: CDRN)
Record Dates: First submitted 2015-03-30; First posted 2015-04-03 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the PaTH Network IPF Clinician-Patient Partnership Cohort is to use clinical data from electronic health records (EHR) and patient reported outcomes (PRO) to answer questions of clinical importance to patients with Idiopathic Pulmonary Fibrosis, providers, and other stakeholders.

DETAILED DESCRIPTION:
The primary objective is to create the PaTH Network IPF Clinician-Patient Partnership Cohort, which will allow the conduct of patient-centered observational studies on IPF across the multiple institutions (Hershey Penn State, University of Pittsburgh, Temple University) of the PaTH network. Creating the IPF Clinician-Patient Partnership Cohort will involve:

1. Recruiting patients with IPF to participate in the PaTH Network IPF Clinician-Patient Partnership Cohort
2. Administering surveys to the IPF Clinician-Patient Partnership Cohort approximately every 3 months to collect patient reported outcomes (PROs)
3. Merging individual patient health record data into the IPF Clinician-Patient Partnership Cohort database
4. Tracking whether the patient participant has biospecimens in a PaTH site biorepository and prepare for possible sharing of biospecimens in future studies.
5. Determining if an automated procedure for identifying duplicate patients across PaTH institutions without the use of protected health information (PHI) is valid compared to a manual matching procedure using PHI.
6. Identifying potential participants for future research studies.

The secondary objectives are to use the PaTH Network IPF Clinician-Patient Partnership Cohort to answer patient-centered research questions including:

1. What is the prevalence of gastroesophageal reflux disease (GERD) in IPF, and what effect does GERD and its treatment have on IPF disease progression, quality of life, and survival?
2. What is the association of oxygen use with survival, quality of life, exercise tolerance, neurocognitive function, and dyspnea?
3. How often do IPF patients have advance directives, how often are advance directives documented in the electronic health record, and does having an advance directive influence how/where IPF patients die, their health care utilization, satisfaction with care, and quality of life?

ELIGIBILITY:
Inclusion Criteria:

* The target study population is adults identified as having IPF (through the PaTH IPF computable phenotype algorithm or a local IPF registry).

Exclusion Criteria:

* Age <18 years
* Deceased
* Not proficient in English
* Has not had at least one outpatient encounter in the past 18 months at the PaTH health system's pulmonary specialty clinic through which they are recruited
* Lung transplant
* Already enrolled in the PaTH Clinician-Patient Partnership Cohort at another PaTH institution

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population is adults with IPF who receive health care at one of the PaTH Network institutions.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Create PaTH Network IPF Clinician-Patient Partnership Cohort | 18 months
  Create the PaTH Network IPF Clinician-Patient Partnership Cohort, which will allow the conduct of patient-centered observational studies on IPF across the multiple institutions (Hershey Penn State, University of Pittsburgh, Temple University) of the PaTH network.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen McTigue, MD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - Johns Hopkins University, Baltimore, Maryland
  - Jody McCullough, Hershey, Pennsylvania
  - Anuradha Paranjape, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah